CLINICAL TRIAL: NCT05986201
Title: Assessment of Long-term Effects of Intraoperative Use of a Carrier-bound Fibrin Sealant (TachoSil®). We Had to Continue to Use it?
Brief Title: Assessment of Long-term Effects of Tachosil
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Isidoro Di Carlo, MD, PhD, FACS, Professor, University of Catania
Other Study IDs: IDC-003
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fibrin Sealant; Haemostasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- 40 patients: There were 33 (82.5%) males and 7 (17.5%) females aged 32-87 years, with a mean age of 67.8 years.
  Interventions: Device: TachoSil®

INTERVENTIONS:
Device: TachoSil® — TachoSil®, a carrier-bound fibrin sealant (CBFS), is a haemostatic tissue sealant composed of a collagen sponge, made from horse tendons, coated on one side with dried human fibrinogen and human thrombin.
  Other Names: haemostatic tissue sealant; carrier-bound fibrin sealant

SUMMARY:
This study aimed to analyse the long-term effects of a carrier-bound fibrin sealant (CBFS) after abdominal surgery by following up patients years after application.

ELIGIBILITY:
Inclusion Criteria:

* type of surgery, indication for surgery, type of disease

Exclusion Criteria:

* dead patients, not available on call.

Ages: 32 Years to 87 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There were 33 (82.5%) males and 7 (17.5%) females aged 32-87 years, with a mean age of 67.8 years.
  The indications for surgery were hepatocellular carcinoma 23 (57.5%), hydatid cyst 3 (7.5%), hepatic adenoma 1 (2.5%), hepatic trauma 2 (5.0%), cholecystitis 2 (5.0%), 3 (7.5%), splenic rupture or bleeding for trauma 1 (2.5%), neuroendocrine tumour and trauma of the pancreas 1 (2.5%), peptic gastric ulcer 3 (7.5%), and colon cancer 1 (2.5%).
  There were 29 hepatic surgical procedures: 4 left lobectomies, 2 right hepatectomies, 9 segmentectomies, 2 bi-segmentectomies, 8 limited resections, and 1 enucleation following the Couinaud classification (23); 2 partial cystopericistectomies, 1 simple suture of the traumatic lobe of the liver after biliary check; 2 cholecystectomies, 3 total splenectomies, 1 enucleation of tumour of the tail of the pancreas, 1 haemostasis of the traumatic tail of the pancreas, 3 sutures of ulcer of the stomach, and 1 colon cancer resection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
fibrotic reaction | 10 years
  The evaluation focused on individuation of the area treated with CBFS, comprehensive analysis of the dimensions of the area treated if visible, and evolution, focusing on the presence of fibrosis, sclerosis, collections, cysts, or pseudocysts. The formation of a fibrotic reaction was related to the presence of residual tissue on CT during follow-up.